CLINICAL TRIAL: NCT04083261
Title: An Observational, Population-Based Study of Pharmacogenetic Variation to Identify Genetic Factors That May Affect the Efficacy and Safety of Medical Marijuana
Brief Title: Pharmacogenetic Variation: Factors That May Affect the Efficacy and Safety of Medical Marijuana
Status: Completed | Type: Observational
Sponsor: Columbia Care Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB Tracking Number: 20190945
Record Dates: First submitted 2019-08-27; First posted 2019-09-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: New York Medical Marijuana Program Qualifying Conditions
Keywords: Medical cannabis; Medical marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High daily dose users: Total Cannabinoid Daily Dose greater than 50 mg
  Interventions: Other: DNA Genotek Oragene 600
- Control: Users that represent the median dose between "high daily dose users" and "low daily dose users" taking between 11-21 mg
  Interventions: Other: DNA Genotek Oragene 600
- Low daily dose users: Total Cannabinoid Daily Dose less than 10 mg
  Interventions: Other: DNA Genotek Oragene 600

INTERVENTIONS:
Other: DNA Genotek Oragene 600 — Saliva-based DNA sample collection kit

SUMMARY:
The primary purpose of this research is to identify genetic factors that may affect the efficacy and safety of medical marijuana, regardless of condition. The pharmacogenomics test detects DNA variants, which may affect the way drugs work and are metabolized in the body and/or detect potential side effects.

DETAILED DESCRIPTION:
This observational, population-based study will examine genetic differences between ultra-rapid, intermediate and poor metabolizers of various formulations of Columbia Care's medical cannabis products in order to identify genetic factors that may affect the efficacy and safety of medical marijuana, regardless of condition. The goal of the research is to establish relationships between cannabis consumers, cannabinoids, and consumer outcomes. The study is expected to enroll 150 subjects across three cohorts, high daily dose users (poor metabolizers) that take more than 50 mg of cannabinoids daily (n=50), low daily dose users (ultra-rapid metabolizers) that take less than 10 mg of cannabinoids daily (n=50), and a control group (intermediate metabolizers) that represents the median daily dose user taking between 11-21 mg of cannabinoids daily (n=50).

Columbia Care Inc. has identified trends amongst its medical cannabis users suggesting that there are some patients who are "high daily dose users" and others who are "low daily dose users", with both groups assumed to have similar satisfaction with the products. The complexity of the endocannabinoid system combined with individual genetic predisposition and gene-environment interactions likely result in the variation in response seen with cannabinoid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18 and older
* Currently obtaining medical marijuana products from Columbia Care LLC
* Willing to participate and consent to a DNA analysis
* Purchased product from Columbia Care for three consecutive encounters spanning a 6-month period

Exclusion Criteria:

* Unwillingness to participate and consent to a DNA analysis
* Unwillingness to answer a survey/questionnaire on patient satisfaction as related to product efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the Columbia Care database (prescription fills/refills and invoice data) and stratified into 3 groups, with n=50 participants in each cohort (total N=150).
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Identification of genetic factors | Day 1
  Saliva-based DNA sample will be tested for known genes (e.g., the cytochrome P-450 superfamily)

SECONDARY OUTCOMES:
Satisfaction with therapy and adverse effects: survey | Day 1
  Survey tool will examine patient satisfaction with current dose as a covariate and evaluate adverse outcomes (e.g., mental health indications, reported unintended effects) based on varying doses and mode of exposure of cannabis within our analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Mazanet, MD, Principal Investigator — Columbia Care Inc.
Locations (1):
- Columbia Care New York Dispensary, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No